CLINICAL TRIAL: NCT02573597
Title: Programmed Intermittent Epidural Bolus (PIEB) Compared to Continuous Epidural Infusion (CEI) Relative Efficacy and Mechanism of Efficacy For Labor Anlagesia: A Minimal Local Analgesic Concentration (MLAC) Study
Brief Title: PIEB vs CEI for Labor Analgesia: An MLAC Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: Stanford University (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Brendan Carvalho, Chief, Division of Obstetric Anesthesia Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 34734
Record Dates: First submitted 2015-09-25; First posted 2015-10-12 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy
MeSH Terms: interventions — Bupivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A Group 1 (Active Comparator): CEI bupivacaine and CEI sufentanil
  Interventions: Drug: Bupivacaine; Drug: Sufentanil
- Part A Group 2 (Active Comparator): PIEB bupivacaine and PIEB sufentanil
  Interventions: Drug: Bupivacaine; Drug: Sufentanil
- Part B Group 3 (Active Comparator): CEI bupivacaine and PIEB sufentanil
  Interventions: Drug: Bupivacaine; Drug: Sufentanil
- Part B Group 4 (Active Comparator): PIEB bupivacaine and CEI sufentanil
  Interventions: Drug: Bupivacaine; Drug: Sufentanil

INTERVENTIONS:
Drug: Bupivacaine — Continuous or bolus administration
  Other Names: marcaine
Drug: Sufentanil — Continuous or bolus administration
  Other Names: sufenta

SUMMARY:
Utilizing a 'minimal local analgesic concentration (MLAC) study' design to first determine the relative potency of Programmed Intermittent Epidural Bolus (PIEB) compared to Continuous Epidural Infusion (CEI) and secondly to determine the mechanism to explain the potential PIEB efficacy advantage.

DETAILED DESCRIPTION:
Pregnant women who present to Labor and Delivery for an anticipated vaginal delivery will be identified as potential participants based on inclusion/exclusion criteria and their desire for labor epidural analgesia. Once identified, interested candidates will be fully informed of the study procedures, have all questions answered, and informed consent obtained. Pregnant participants will receive a labor epidural upon the patient's request and dosed per protocol to adequate analgesic level.

Patients will be randomized into 1 of 4 groups. Either group I or II in Study Part A and group III or IV in Study Part B in a double-blinded design. Each study part will run in parallel and independently.

Each group will have a varying concentration of bupivicaine infusion; continuous or intermittent bolus administration. In addition each group will have continuous or intermittent bolus administration of sufentanil. These concentrations and forms of administration will be blinded to both the patient and study administrator.

Each epidural infusion concentration and continuous or bolus administration will be determined to be a success or failure based on analgesic scores. The investigators' primary outcome will be the minimal local anesthetic concentration of the final participants in each respective group upon study completion.

DATA SAFETY MONITORING PLAN will follow standard of clinical care. Any adverse events will be reported to the PI and necessary adjustments to the protocol will be immediately instituted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II, Nulliparous and Multiparous, Spontaneous/Induced/Augmented Labor, Early active labor (cervix <5 cm (if known)), Pain (VPS) > 3, 18-45 years of age

Exclusion Criteria:

* <37 weeks gestation, H/o Cesarean Section, Multiple Gestation, Pre-eclampsia, Narcotics within 3 hours prior to labor epidural placement, Chronic Pain (as defined by chronic opiate consumption), Women who are participating in another study that will impact protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MBBCh, MDCH, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

REFERENCES:
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Ginosar Y, Columb MO, Cohen SE, Mirikatani E, Tingle MS, Ratner EF, Angst MS, Riley ET. The site of action of epidural fentanyl infusions in the presence of local anesthetics: a minimum local analgesic concentration infusion study in nulliparous labor. Anesth Analg. 2003 Nov;97(5):1439-1445. doi: 10.1213/01.ANE.0000081792.84877.A2. PMID 14570662

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who met the protocol-specified "reject" criteria were censored (had no subsequent outcome measure data collected and were not considered analyzable for outcome measures) and were considered to have completed the study. Upon reject, catheter management was at discretion of anesthesia care provider.
Period: Overall Study
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Started | 8 | 6 | 9 | 8
Met Reject Critera | 4 | 1 | 3 | 2
Analyzable Data Set | 4 | 5 | 6 | 6
Completed | 8 | 6 | 9 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4 | Total
Number analyzed (Participants) | 8 | 6 | 9 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (7.2) | 30 (5.7) | 33.1 (6.1) | 30.6 (6.8) | 32.0 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 9 | 8 | 31
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 1 | 5 | 3 | 14
  Hispanic | 2 | 1 | 1 | 2 | 6
  Asian | 1 | 4 | 2 | 2 | 9
  American Indian/Alaska Native | 0 | 0 | 0 | 1 | 1
  Not reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 9 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Minimum Local Analgesic Concentration (MLAC) of the Final Participants in Each Respective Group at Study Completion
Description: The mean concentration of Bupivacaine in patients who have success or failure outcome were compared between groups.
Time Frame: From initial epidural bolus to delivery (up to approximately 16 hours)
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Mean (Standard Deviation); unit: % mg/ml
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
% mg/ml | 0.06 (0.008) | 0.06 (0.007) | 0.075 (0.010) | 0.072 (0.008)

2. Secondary Outcome: Time to First Clinician Rescue Analgesia Request (From Initial Epidural Dose)
Description: The time to first clinician rescue analgesia request in patients who have success or failure outcome were compared between groups.
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
hours | 4.3 (1.7) | 5.3 (1.2) | 7.5 (5.2) | 4.8 (3.0)

3. Secondary Outcome: Numerical Verbal Pain Scores
Description: The initial pain score (VAS 0-10 scale with 0 means no pain and 10 means max pain) in patients who have success or failure outcome were compared between groups.
Time Frame: Patients were assessed once between initial epidural bolus to delivery (up to 16 hours following initial bolus)
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
score on a scale | 6.3 (1.0) | 8.4 (0.9) | 7.7 (2.1) | 8.2 (1.0)

4. Secondary Outcome: Patient Satisfaction With Labor Analgesia
Description: 0-100% (0 means least satisfaction and 100 means most satisfaction)
Time Frame: Participants were assessed once from initial epidural bolus to delivery (up to approximately 16 hours)
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
score on a scale | 97.3 (4.9) | 97.6 (4.3) | 99.2 (2.0) | 96.7 (5.2)

5. Secondary Outcome: Labor Outcome (Spontaneous, Assisted, Cesarean)
Description: Labor outcome in patients who have success or failure outcome were compared between groups.
Time Frame: At the time of delivery
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
Participants
  Spontaneous | 3 | 3 | 4 | 6
  C-section | 1 | 2 | 2 | 0

6. Secondary Outcome: Number of Participants Requiring Treatment for Pruritus, Nausea and Vomiting, or Hypotension
Description: Number of Participants Requiring Treatment for pruritus, nausea and vomiting, and hypotension were reported.
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
Participants | 0 | 0 | 2 | 3

7. Secondary Outcome: Number of Participants With Maternal Nausea/Vomiting
Description: yes/no.
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
Participants | 0 | 0 | 0 | 2

8. Secondary Outcome: Protocol Success or Failure
Description: Success - No supplemental analgesia request until vaginal exam c/w 8 cm dilation or more -> 0.01% w/v reduction in subsequent participant's local anesthetic.
  Failure - Supplemental analgesia request c vaginal exam c/w less than 8 cm dilatation ->0.01% w/v increase in subsequent LA infusion.
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Population: Analyzable data set (did not meet the protocol-specified "reject" criteria).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
Number analyzed (Participants) | 4 | 5 | 6 | 6
Participants
  Success | 1 | 3 | 2 | 2
  Failure | 3 | 2 | 4 | 4

9. Other Pre Specified Outcome: Maternal Pruritis
Description: scale from from 0-10
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Motor Weakness
Description: Straight leg lift, yes/no
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number and Total Dose of Clinician Rescue Boluses
Time Frame: From initial epidural bolus to approximately 6-12 hours following delivery
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Total CEI and PIEB Local Anesthetic and Opioid Use
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Requests to Turn Epidural Down or Stop Infusion.
Description: yes/no
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Duration of Epidural Analgesia
Time Frame: From initial epidural bolus to delivery (up to 16 hours following initial bolus)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From initial epidural bolus to delivery (up to approximately 16 hours)
Arm/Group | Part A Group 1 | Part A Group 2 | Part B Group 3 | Part B Group 4
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/9 | 0/8

LIMITATIONS AND CAVEATS:
This study did not meet its planned enrollment and did not achieve power for the intended analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT02573597/Prot_SAP_000.pdf